CLINICAL TRIAL: NCT06467474
Title: Psychoeducation for Major Depressive Disorder: Development and Evaluation of Effectiveness
Brief Title: Psychoeducational Group for Depression
Acronym: PEG-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ricardo Alberto Moreno, M.D., Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Ricardo Alberto Moreno, M.D., Ph.D., PhD, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 76212623.1.0000.0068
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder (MDD
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Group (Experimental): Participants will receive treatment as usual (TAU) associated with the psychoeducational program.
  Interventions: Behavioral: PEG-D program; Drug: TAU
- Control Group (Active Comparator): The usual treatment will consist of outpatient follow-up for a period of twelve months.
  Interventions: Drug: TAU

INTERVENTIONS:
Behavioral: PEG-D program — PEG-D will be carried out in person, open format, for six consecutive weeks lasting 90 minutes each. An approximate group of 6 to 10 participants will be led by a team of experienced psychologists and psychiatrists. Each group will have a main therapist and a co-therapist to ensure effective support and guidance for participants. Before the start of the group, participants received a booklet containing the content of the sessions.
  Arms: Clinical Group
Drug: TAU — The treatment will start with Sertraline (SSRI) - doses of 50 mg and adjusting as necessary according to the patient's profile. After 8 weeks, if the patient experiences remission, they will continue on monotherapy with Sertraline. In case of relapse Bupropion, Quetiapine, Lithium or Aripiprazole might be add-on. In this case, add-on medications will be determined according to the patient profile, by the clinician. If there is a response above 25% of the symptoms, but without remission, the patient will proceed to augmentation with the aforementioned medications and if there is no improvement of at least 25%, the patient will be considered drop-out. Associations with Lorazepam if necessary will be allowed in any phase of the study.

SUMMARY:
The study aims to investigate the efficacy of a psychoeducational program as an adjunctive treatment for depression. The study will involve 338 patients diagnosed with Major Depressive Disorder (MDD) of moderate severity. Participants will be randomly assigned to receive either Treatment as usual (TAU) alone or TAU plus the psychoeducational program. The program consists of six weekly group sessions covering information and techniques for coping with depression. Primary outcomes include a reduction in depressive symptoms measured by the Beck Depression Inventory-II (BDI-II) and increased knowledge of depression. Secondary outcomes include improvements in functionality and quality of life. The study aims to provide insights into the effectiveness of psychoeducation in improving outcomes for individuals with depression

ELIGIBILITY:
Inclusion:

* Both sexes;
* Ages between 18 and 65 years old;
* Diagnosis of Major Depressive Disorder (MDD) made by a clinician according to Diagnostic Statistical Manual criteria-5-Text Revised (DSM-5-TR)
* Patients with Hamilton Depressive Rating Scale-17 items (HDRS-17) scores 14-23;
* Informed and signed consent form.

Exclusion:

* Unstable serious clinical or neurological diseases;
* Postpartum depression or other types of depressive disorders (disruptive mood dysregulation disorder, pre-menstrual, substance/medication-induced depressive disorder, depressive disorder due to another medical condition, another disorder specified depressive disorder and unspecified depressive disorder);
* Other psychiatric disorders;
* Patients with active psychotic symptoms;
* Suicidality risks
* Patients already undergoing any other psychological treatment for MDD;

Discontinuation:

* More than two absences during treatment;
* Those who miss more than two sessions/consultations, whether medical treatment or the psychoeducational program;
* Non-response to the use of Sertraline over the initial eight weeks; Presence of hypomanic symptoms at any time during treatment (Young <7)

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 338 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge level | Time: baseline, post 6 weeks and 12 months.
  Learning quiz: Comprising of open and closed questions questions, it was designed to evaluate participants' level of knowledge regarding depression
Depressive levels | Baseline, post 6 weeks, 3, 6 and 12 months.
  Beck Depression Inventory-BDI-II. It consists of 21 items and measures the intensity of depression in the last 14 days. The instrument has 21 items, and the higher the score, the greater the intensity of depression.

SECONDARY OUTCOMES:
Depressive Thoughts | Baseline, post 6 weeks, 3, 6 and 12 months
  Depressive Thoughts Scale (EPD): The instrument has 26 items, divided into two factors, the first being low self-esteem/hopelessness, with 16 items referring to the subject's negative perception of themselves and their future perspectives and the second on functionality in relationships, with 10 items on the positive evaluation that the subject presents about their relationship with others and how they evaluate the support they receive.
Avoidance behaviors | Baseline, post 6 weeks, 3, 6 and 12 months.
  Cognitive Behavioral Avoidance Scale (CBAS): The instrument assesses typical avoidance styles of depressed people and has 31 items, divided into four factors, namely: Behavioral/Social (8 items), Non-Social Behavioral (6 items), Social Cognitive (7 items) and Non-Social Cognitive ( 10 items).
Functionality | Baseline, post 6 weeks, 3, 6 and 12 months.
  Global Functioning Ranting Scale (GAF): The GAF is a functioning assessment scale that ranges from 0 to 100, with higher scores indicative of higher levels of functioning. The Clinical Global Impression Scale (CGI) will also be used, a general summary measure determined by the physician that takes into account all available information, including knowledge of the patient's history and the impact of symptoms on the patient's functional capacity, with measures ranging from 1 (much better) to 7 (much worse).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry - Faculty of Medicine from University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Carneiro AM, Silva SLT, Fernandes FDS, Barretto JR, de Brito TR, Moreno LH, Pimentel FC, Jorge BA, Dos Santos LA, Fernandes Ramos MR, Moreno RA. Psychoeducation Group for Depression (PEG-D): Study protocol for a prospective, randomized, single-blind, crossover trial. PLoS One. 2025 Aug 8;20(8):e0329006. doi: 10.1371/journal.pone.0329006. eCollection 2025. PMID 40779501